CLINICAL TRIAL: NCT06169683
Title: Evaluation of Daily- and Extended-wear Hearing Instruments
Brief Title: Lyric4 Outcomes Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-6569
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hearing Loss
Keywords: hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experienced Lyric Users (Experimental): This cohort of participants is required to have Lyric hearing instrument experience, and they will be asked to wear Lyric for the duration of the study period and report on their experience.
  Interventions: Device: Lyric4

INTERVENTIONS:
Device: Lyric4 — Lyric4 Hearing instrument use

SUMMARY:
The goal of this clinical investigation is to obtain feedback on Lyric4 device updates within a cohort of experienced adult Lyric hearing instrument users. The main question it aims to answer is:

• Do device updates cause a change in Lyric patient experience?

Participants will be asked to complete questionnaires about their past experience with Lyric, as well as their experience with Lyric during the study period. They will also be asked to undergo aided audiometric testing with Lyric devices.

ELIGIBILITY:
Inclusion Criteria:

* Experience with Lyric hearing instruments
* Willingness to travel to the study site and complete study procedures
* Adults, age 18 or older
* Fluency with English (written/spoken)

Exclusion Criteria:

* No Lyric hearing instrument experience
* Ear health issues preventing Lyric fitting or requiring medical clearance prior to fitting
* Difficulty reading when corrected for vision loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Aided Audiometric Testing | From enrollment to the end of the study period, approximately one month.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sonova Silicon Valley, Fremont, California
  - Triangle Hearing Services, Cary, North Carolina

IPD SHARING:
Plan to Share IPD: No